CLINICAL TRIAL: NCT03665805
Title: Neuromuscular Monitoring, Reversal of Block and Postoperative Residual Curarization: the Situation in 2018
Brief Title: Postoperative Residual Curarization in 2018
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Guy CAMMU, Staff Anesthesiologist, Onze Lieve Vrouw Hospital
Other Study IDs: LKGC2018
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Residual Curarization
Keywords: Muscle Relaxation
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: neuromuscular transmission monitoring — The acceleromyographic responses of the adductor pollicis muscle as percent of the train-of-four (TOF%) on stimulation of the ulnar nerve by means of the TOFscan neuromuscular transmission monitor (iDMed, Marseille, France).

SUMMARY:
The primary objective of this study is to evaluate the incidence of postoperative residual curarization, as defined by a train-of-four <90%, upon postanaesthesia care unit arrival. Anesthetists tend to use train-of-four monitoring in the operating theatre to interpret muscle tone. Train-of-four monitoring is a widely used term for the peripheral nerve stimulation used in neuromuscular blockade monitoring. Hypothesizing a change in our practice since 2006-2012 (Cammu G, Anesth Analg 2006; 102: 426-9 and Cammu G, Anaesth Intensive Care 2012; 40: 999-1006), residual neuromuscular block as well as the use of intraoperative neuromuscular transmission monitoring and reversal of neuromuscular blocking agents will again be prospectively evaluated in 2018. The present study aims to compare these three periods (2006-2012-2018) in terms of management of neuromuscular block in the operating room and to look for a relationship with the incidence of postoperative residual curarization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Informed consent signed;
* Admission for elective surgery;
* Administration of non-depolarizing neuromuscular blocking agents during surgery;
* Tracheal intubation

Exclusion Criteria:

* Evidence of renal, hepatic, metabolic, and/or neuromuscular disorders
* Ejection fraction <20%
* Admission for emergency surgery; or cardiothoracic surgery
* Reoperation during the same hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 600 surgical patients (the first 600 inpatients and outpatients scheduled for anesthesia during the study period who meet the study criteria).
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative residual curarisation | Immediately after the patients' arrival in the post-anesthesia care unit (<5 min after arrival), two consecutive neuromuscular transmission measurements (separated by 15 s) will be obtained, and the average of the 2 values will be recorded.
  Incidence of postoperative residual curarisation defined by a train-of-four (TOF) ratio < 0,9 at post-anesthesia care unit arrival

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Hospital, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cammu G, De Witte J, De Veylder J, Byttebier G, Vandeput D, Foubert L, Vandenbroucke G, Deloof T. Postoperative residual paralysis in outpatients versus inpatients. Anesth Analg. 2006 Feb;102(2):426-9. doi: 10.1213/01.ane.0000195543.61123.1f. PMID 16428537
- [Background] Cammu GV, Smet V, De Jongh K, Vandeput D. A prospective, observational study comparing postoperative residual curarisation and early adverse respiratory events in patients reversed with neostigmine or sugammadex or after apparent spontaneous recovery. Anaesth Intensive Care. 2012 Nov;40(6):999-1006. doi: 10.1177/0310057X1204000611. PMID 23194209